CLINICAL TRIAL: NCT05138237
Title: Evaluation of Different Modalities (Surgery and Endoscopy) in Management of Indeterminate Lower Common Bile Duct Stricture
Brief Title: Evaluation of (Surgery and Endoscopy) in Management of Indeterminate Common Bile Duct Stricture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mohamed Elsayed Abdelaal, assistant lecturer of general surgery sohag faculty of medicine, Sohag University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: Soh-Med-21-10-30
Record Dates: First submitted 2021-10-15; First posted 2021-11-30 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: Indeterminate Common Bile Duct Stricture
Keywords: common bile duct stricture \ indeterminate
MeSH Terms: interventions — Endoscopy; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- benign stricture (Active Comparator): no of cases suspected to be benign by using the diagnostic tools "imaging , laboratory investigations , ERCP ,brushing ,cytology or histopathology"
  Interventions: Procedure: endoscopy or surgery
- malignant stricture (Active Comparator): no of cases suspected to be malignant by using the diagnostic tools "imaging , laboratory investigations , ERCP ,brushing ,cytology or histopathology"
  Interventions: Procedure: endoscopy or surgery

INTERVENTIONS:
Procedure: endoscopy or surgery — we choose the proper intervention "surgery or endoscopy" for management of the indeterminate common bile duct stricture according to its nature benign or malignant

SUMMARY:
Evaluate the lower indeterminate CBD strictures trying to reach possible diagnosis by all available methods i.e brush cytology ,bile aspirate cytology , tissue biopsy ,imaging studies and laboratory work up then treatment of the patient either endoscopically or surgically according to the etiology.

DETAILED DESCRIPTION:
Aim of the work Evaluate the lower indeterminate CBD strictures trying to reach possible diagnosis by all available methods i.e brush cytology ,bile aspirate cytology , tissue biopsy ,imaging studies and laboratory work up then treatment of the patient either endoscopically or surgically according to the etiology.

Approvals and consents This study will be done after obtaining approval by the medical ethics committee of sohag faculty of medicine.A written informed consent will be obtained from all participants before being enrolled in the study and prior to performing the procedure .the study will be registered in www.clinicaltrials.gov .

Clinical presentation The common presentation is one or more of Charcot's triad ;Jaundice ,Fever and Pain with itching and dark urine and pale clay stool Also the patient may be presented by Pain in the upper right side of the abdomen (biliary pain) ,nausea and vomiting .

By examination yellowish discoloration of skin and sclera and mucous membrane , and itching marks.

Accidental diagnosis of indeterminate stricture may be discovered in asymptomatic patient during imaging study (MRCP , US), or during ERCP for any other cause i.e common bile duct stone after stone extraction accidently a distal CBD stricture

Laboratory Assessment:

routine investigations: CBC , coagulation profile, kidney function liver function : total \direct bilirubin ductal enzymes i.e Alkaline phosphatase ,gamma glutamyl transferase GGT, 5-nucleotidase.

Tumour markers for cases suspected to be malignant and old aged patients: CA19.9 ,AFP (alpha-fetoprotein) ,and CEA (carcino-embryonic antigen)

Imaging study:

imaging US ,MRCP routinely done for all cases Triphasic CT abdomen and pelvis if needed

Endoscopic Technique ERCP done routinely for all cases of indeterminate lower common bile duct stricture to help reaching diagnosis. The patient is positioned in prone position with slight elevation of the right shoulder to improve the orientation . the anesthesia will be propofol intravenous as sedation with monitoring of the vital signs. introduction of the scope till facing the papilla, iv injection of hyoscine butyl bromide will decrease duodenal motility and allow easy successful cannulation followed by Sphincterotomy .

By injection of bilograffin contrast The radiological configuration of the stricture in the cholangiogram is either irregular with shouldering suggesting malignancy or smooth tapered nature suggesting benign stricture . Also the cholangiogram will evaluate the stricture if it is affecting long or short CBD segment .After cannulation and sphincterotomy a guide wire will be introduced in the biliary passage.

Biopsy either punch biopsy if there's papillary overgrowth will be taken by biopsy forceps or core biopsy from the stricture itself will be taken during ERCP and sent for histopathology.

Brush cytology After confirmation of the Presence of CBD stricture which is distal in position "beyond cystic duct " by the cholangiography , a double lumen cytology brush will passed into bile duct beyond the stricture over a guide wire .

The brush will be pushed into the stricture as this region will be abraded by rapid forward and back movement of the brush more than 5-6 times . finally the brush will be pulled in the catheter sheath again, and both the brush and the sheath will be removed from the endoscope as a unit . The samples will be divided into two parts one for CCE "Conventional cytology evaluation" and the other for Digital image Analysis( DNA histogram) examination .

Bile Aspirate Cytology In some cases bile aspirate will be done before injecting the contrast in the bile duct ,The sample will be centrifuged and the sediment will be used to perform CCE and DIA.

From each patient ,two samples obtained one of them will be fixed immediately in 2 ml of phosphate buffer solution and will be sent for DIA. The other sample will be sent to pathology center at Sohag University for conventional cytology evaluation CCE.

Samples will be preserved in 75 % alcohol .Centrifugation will be done for 30 minutes and the sediment will be directly smeared onto one or more glass slides ,fixed using alcohol based fixative and stained with Papanicolaou stain .

Cells will be labelled as malignant based on the following criteria; loss of honeycombing ,loss of polarity ,increased nuclear size ,increased nuclear cytoplasmic ratio, chromatin clumping, nuclear molding and presence of dirty ,necrotic or bloody background .Absence of such features will be consistent with benign nature.

The cytometric estimation of DNA aberration is commonly expressed as DNA index (DNA-I). This index is a measure of DNA aneuploidy or abnormal DNA content . DNA-I of 1.0 represents a normal diploid DNA content .

DNA ploidy analysis will be done by BD cycle test TM plus DNA kit (BD ;san joe ,CA95131 ,USA). DNA histogram will be generated for ploidy analysis automatically by plotting individual nuclear DNA content against number of nuclei.

Firstly ,five samples will taken from five patients with benign biliary obstruction other than stricture "calcular obstructive jaundice) to assign DNA histogram and DNA-I of normal biliary cells. Results of DNA-I will placed into 1 of 4 categories, which identified nuclei with DNA indices between 0.95 and 1.05 (diploid), 1.06 and 1.89(aneuploid or S phase), 1.90 and 2.10 (tetraploid), or greater than 2.10 (hypertetraploid). Aneuploid ,tetraploid ,and hypertetraploid are considered positive for malignancy.

Dilatation and stenting Therapeutic role of ERCP is very important ,After diagnosing the stricture frequent dilatation by disposable soehendra biliary dilatation catheter will be done or by balloon dilatation.Then stent insertion will be done and upgraded later on according to the stricture .Benign strictures are more amenable for endoscopic dilatation by ERCP in one or more than one ERCP sessions .

Malignant stricture which is inoperable managed endoscopically with ERCP and metal stenting.

EUS EUS used in some cases to determine the nature of stricture and its criteria if it is regular smooth or irregular infiltrative to the surroundings or it is compressing extraluminal mass lesion. EUS guided FNA cytology will be done from any suspicious lesions .

Surgical technique

Strictures proved to be benign will undergo endoscopy but surgery is mandatory in case of bad patient compliance for endoscopy; the operation will be shunt operation ( bilio-enteric anastomosis) in the form of :

* proximal choledocho-duodenostomy (side to side)
* proximal choledocho-jejunostomy (side to side)
* proximal choledocho-duodenostomy (end to side) with excision of the strictured segment .
* proximal choledocho-jejunostomy (end to side) with excision of the strictured segment.

Strictures proved to be malignant if operable will undergo:

* Excision of the stricture with safety margin + shunt operation (bilio-enteric anastomosis end to side) + regional draining LNs block dissection.
* Pancreatico-duodenectomy (Whipple's operation) Strictures proved to be malignant if inoperable will undergo: endoscopy

Follow up Follow up of the patients will be for 6-9 months post treatment . those with lower common bile duct (CBD strictures managed endoscopically will undergo ERCP sessions for stent upgrading and re-evaluation of the stricture .

Patients will be followed up Clinically or by imaging studies (US, MRCP , CT abdomen) if needed to detect the progression of the disease .

Statistical Analysis Data will be collected in preformed data collection from prior to being entered in the spread sheet. Statistical analysis will be performed using the statistical package for social science (SPSS).continuous variables will be expressed as mean and standard deviation (normal distributed data) or median and range (not normal distributed data) while categorical data expressed as numbers and percentages.

Chi square test will be used to compare the nominal data while continuous data will be compared by student t test(normally distributed data) and Mann Whitney test (not normally distributed data).

ELIGIBILITY:
Inclusion Criteria:

* both sex
* above age of 20 years old
* patients presented with jaundice , pain and fever due to lower common bile duct stricture evident by abdominal imaging (Abdominal US ,MRCP) and confirmed by endoscopic retrograde cholangiopancreatography ( ERCP)
* patients presented to sohag university hospital.

Exclusion Criteria:

* Already diagnosed lower CBD strictures i.e known cause like visible pancreatic mass with visible metastasis or common bile duct stones.
* Coagulopathy INR more than 1.5 or thrombocytopenia platelet less than 50,000/ml.
* Proximal common bile duct stricture "above level of cystic duct".

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-08-01 (Estimated); Study Completion 2023-02-01 (Estimated)

PRIMARY OUTCOMES:
number of patients who are successfully treated of CBD strictures by endoscopy or by surgery | follow up of the patient for 6 - 9 months
  dilatation or resection and shunt operation of CBD strictures allow continuity of the biliary system with good bile drainage
reach a proper algorithm or scheme for management of the CBD stricture | follow up of the patient for 6 - 9 months
  reach a proper algorithm or scheme to help in diagnosis of CBD strictures also, choose the proper method for treatment according to the nature and criteria of the CBD stricture

SECONDARY OUTCOMES:
number of patients diagnosed by each method to measure accuracy and sensitivity of each method used in the study in diagnosis of biliary strictures | follow up of the patient for 6 - 9 months
  comparing results with each method of diagnosis of CBD stricture

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag Faculty of Medicine, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided